CLINICAL TRIAL: NCT00726830
Title: A Randomized Comparison of Oral Methadone as a "First-Switch" Opioid Versus Opioid Switching Between Sustained-Release Morphine and Oxycodone for Oncology-Hematology Outpatients With Pain Management Problems: The "Simply Rotate" Study
Brief Title: Methadone, Morphine, or Oxycodone in Treating Pain in Patients With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-0791; MDA-2007-0791; CDR0000598283 (Other: NCI Identifier)
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Results first posted 2012-12-06 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Brain and Central Nervous System Tumors; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Pain; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: pain; unspecified adult solid tumor, protocol specific; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated hairy cell leukemia; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related lymphoblastic lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; HIV-associated Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; cutaneous B-cell non-Hodgkin lymphoma; Waldenström macroglobulinemia
MeSH Terms: conditions — Central Nervous System Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Pain; Precancerous Conditions; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Waldenstrom Macroglobulinemia | interventions — Methadone; Morphine; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Opioid rotation to oral methadone (Experimental): Participants are switched from their current opioid medication (oxycodone or morphine) to methadone. Participants receive oral methadone 2-3 times daily for 4 weeks.
  Interventions: Drug: methadone hydrochloride
- Arm II: Opioid rotation to another long-acting strong opioid (Experimental): Participants currently receiving oxycodone are switched to sustained-release (SR) morphine. Participants currently receiving morphine are switched to SR oxycodone. Participants receive either oral SR morphine or oxycodone 2-3 times daily for 4 weeks.
  Interventions: Drug: morphine sulfate; Drug: oxycodone hydrochloride

INTERVENTIONS:
Drug: methadone hydrochloride — Given orally
  Other Names: methadone; dolophine; methadose
  Arms: Arm I: Opioid rotation to oral methadone
Drug: morphine sulfate — Given orally
  Arms: Arm II: Opioid rotation to another long-acting strong opioid
Drug: oxycodone hydrochloride — Given orally
  Other Names: oxycodone; ETH-Oxydose; DSC; OxyIR; OxyContin; Roxicodone
  Arms: Arm II: Opioid rotation to another long-acting strong opioid

SUMMARY:
RATIONALE: Methadone, morphine, or oxycodone may help relieve pain caused by cancer. It is not yet known whether methadone is more effective than morphine or oxycodone in treating pain in patients with cancer.

PURPOSE: This randomized clinical trial is studying methadone to see how well it works compared with morphine or oxycodone in treating pain in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the effectiveness of an opioid rotation to oral methadone versus an opioid rotation to another long-acting strong opioid (sustained-release morphine or oxycodone) in controlling pain (i.e., analgesia) in patients with cancer.

Secondary

* To compare the tolerability of an opioid rotation to oral methadone versus an opioid rotation to another long-acting strong opioid (sustained-release morphine or oxycodone).
* To identify a subset of patients most likely to benefit from an opioid rotation to oral methadone, in terms of significant improvement in pain control or opioid tolerability.

OUTLINE: This is a multicenter study. Patients are stratified according to their baseline opioid (morphine vs oxycodone). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients are switched from their current opioid medication (oxycodone or morphine) to methadone. Patients receive oral methadone 2-3 times daily for 4 weeks.
* Arm II: Patients currently receiving oxycodone are switched to sustained-release (SR) morphine. Patients currently receiving morphine are switched to SR oxycodone. Patients receive either oral SR morphine or oxycodone 2-3 times daily for 4 weeks.

Patients are assessed for pain control and complete a symptom questionnaire on days 1, 8, 15, 22, and 28.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Receiving ongoing care in the outpatient medical oncology setting
* Self-reported pain (of any cause) for which long-acting strong opioids (morphine or oxycodone) have been prescribed or administered

  * Oral morphine-equivalent daily dose (MEDD) of existing opioid regimen (long-acting or immediate-release) 40-300 mg/day
* Worst pain score on a scale of 0 (no pain) to 10 (worst pain) of ≥ 5 for ≥ 1 week duration based on verbal self-report AND/OR ≥ 1 persistently bothersome symptom attributed to an opioid side effect (e.g., fatigue, confusion, depressed level of consciousness, memory loss, personality change, anorexia, constipation, dehydration, nausea, vomiting, weight loss, pruritus, urticaria, impotence, reduced libido, and urinary retention or hesitancy)

PATIENT CHARACTERISTICS:

* None of the following conditions that could predispose the patient to prolonged QT interval-associated tachycardia:

  * Serum potassium < 3.0 mg/dL
  * Cocaine abuse within the past 3 months
  * Family history of sudden death
  * Advanced heart failure (ejection fraction < 40% and/or New York Heart Association (NYHA) class III or IV heart disease)
* No known or suspected cognitive impairment that could interfere with adherence to the medication plan or self-report of symptoms and side effects
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy or surgery for local control of cancer or pain palliation
* More than 60 days since prior use of the same long-acting opioid (i.e., the new long-acting opioid) that patient is switching to on the study
* More than 12 weeks since prior methadone therapy
* More than 3 days since prior and no concurrent transdermal fentanyl, oxymorphone, or buprenorphine
* Concurrent systemic anticancer therapy or bisphosphonates allowed provided therapy was initiated ≥ 4 weeks ago
* Concurrent tricyclic antidepressants, Nonsteroidal Antiinflammatory Drugs (NSAIDs), anticonvulsants, or other adjuvant analgesics or psychostimulants allowed provided therapy was initiated ≥ 2 weeks ago

  * Dose expected to remain stable until after the first week of opioid rotation on study
* No concurrent methadone maintenance therapy for opioid addiction
* No concurrent intrathecal infusion of analgesics
* No concurrent antiarrhythmic medications (e.g., amiodarone or quinidine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Fisch, MD, MPH, FACP, Study Chair — M.D. Anderson Cancer Center; James D. Bearden, MD, Study Chair — CCOP - Upstate Carolina
Locations (2):
- United States (2):
  - Palmetto Hematology Oncology, PC at Gibbs Regional Cancer Center, Spartanburg, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 10, 2009 to October 1, 2010. Recruitment occured within University of Texas MD Anderson Cancer Center and Palmetto Hematology Oncology at Gibbs Regional Cancer Center.
Period: Overall Study
Arm/Group | Arm I: Opioid Rotation to Oral Methadone | Arm II: Opioid Rotation to Another Long-acting Strong Opioid
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Opioid Rotation to Oral Methadone | Arm II: Opioid Rotation to Another Long-acting Strong Opioid | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least a 3-point Reduction in Pain Score on the M.D. Anderson Symptom Inventory (MDASI)
Description: MDASI questionnaire completed on days 8, 15, and 22 after enrollment. The 'primary success' is defined as a 3-point reduction in pain score on the MDASI. Scores from baseline and from four weeks later compared using the MDASI average pain intensity on a scale of 0 (no pain) to 10 (worst pain).
Time Frame: 28 days
Population: No Analysis accomplished as there is not sufficient participant data to meet the study end points.
Arm/Group | Arm I: Opioid Rotation to Oral Methadone | Arm II: Opioid Rotation to Another Long-acting Strong Opioid
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With 30% Reduction in Total Summary Score for the Individual Composite Drug Toxicity Score (CDTS) Items
Time Frame: 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 Months
Arm/Group | Arm I: Opioid Rotation to Oral Methadone | Arm II: Opioid Rotation to Another Long-acting Strong Opioid
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No